CLINICAL TRIAL: NCT03223870
Title: Respiratory Rate Accuracy - Healthy Adults
Status: Completed | Type: Observational
Sponsor: Nonin Medical, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: QATP3064
Record Dates: First submitted 2017-07-13; First posted 2017-07-21 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Normal Respiration Patterns
MeSH Terms: interventions — Diagnosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Oximeters: Comparison of respiratory rates with other devices in normal subjects as observational with other pulse oximeters. No treatment of interventions will be performed.
  Interventions: Diagnostic Test: Diagnostic

INTERVENTIONS:
Diagnostic Test: Diagnostic — Diagnostic

SUMMARY:
The objective of this study is to evaluate the Fingertip Respiratory Rate algorithm performance of the Nonin Medical X-100SP pulse oximetry systems with the 8300AA sensors and Onyx 3 fingertip oximeter. There is no treatment or interventions being performed.

DETAILED DESCRIPTION:
1. Start data collection system(s) and allow them to run 15 minutes prior to study start of each subject.
2. Confirm that the subject meets inclusion/exclusion criteria and has signed the current IRB- approved Informed Consent Form
3. Collect Demographic and Anthropometric Data from the subject.
4. Place Pulse Oximetry Sensors
5. Place nasal cannula for capnography recordings
6. A summary of Respiratory rate protocol.

   1. Stage 1: Subject will rest quietly and breathe at a normal comfortable rate for 40 minutes. The start and stop times will be marked on the data collection system.
   2. Stage 2: Immediately after Stage 1 is complete, the subject will start the 25 minute paced breathing protocol which will ramp from 5-45 BPM. A computer program will be used to guide the subject through the stage 2 paced breathing. The start and stop times will be marked on the data collection system.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female
* The subject is of any racial or ethnic group
* The subject is > 30 kg (>66 pounds) in weight (based on measurement)
* The subject has at least one finger with a height of 0.3 - 1.0 inch (7.6 -25.4 mm) (based on measurement)
* The subject is between 18 years and 50 years of age (self-reported)
* The subject has given written informed consent to participate in the study
* The subject is both willing and able to comply with study procedures.

Exclusion Criteria:

* The subject has a BMI greater than 30 (based on weight and height)
* The subject has a history of atrial fibrillation (self-reported)
* The subject has a documented history of frequent premature ventricular contractions (PVCs), defined as >3 per 30 seconds (self-reported)
* The subject has an implanted pacemaker (self-reported)
* The subject has had any relevant injury at the sensor location site (self-reported)
* The subject has deformities or abnormalities that may prevent proper application of the device under test (based on examination)
* The subject has a known respiratory condition (self-reported)
* The subject has a known heart or cardiovascular condition (self-reported)
* The subject is currently pregnant (self-reported)
* The subject is actively trying to get pregnant (self-reported)
* The subject is unwilling or unable to provide written informed consent to participate in the study
* The subject has another health condition which in the opinion of the principal investigator makes him/her unsuitable for testing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A minimum of 30 subjects will be included in this study. The subject selection will be an approximately equal mix of males and females with varying skin tones. At a rate of 3-4 subjects per day, enrollment will take approximately 7-10 days to complete.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Respiratory Rate Accuracy | 3 months
  Values from the test device will be compared to the values from co-oximetry devices

CONTACTS AND LOCATIONS:
Overall Officials: Walter Holbein, Ph.D, Principal Investigator — Nonin Medical, Inc
Locations (1):
- Nonin Medical, Inc., Plymouth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No